CLINICAL TRIAL: NCT04339621
Title: AIH Risk Stratification With Multiparametric MRI
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: EC-88
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Autoimmune Hepatitis
Keywords: Autoimmune hepatitis; LiverMultiscan; MRI; Liver Biopsy
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Treatment Naive: 20 patients with AIH will be recruited that will be treatment naive at the time of recruitment.
  Interventions: Device: LiverMultiscan
- Treatment cessation review: 77 AIH patients will be recruited who will have been on treatment for the past 18-24 months and will be coming in to meet their physician to review treatment cessation options
  Interventions: Device: LiverMultiscan

INTERVENTIONS:
Device: LiverMultiscan — The LiverMultiscan is a quick 15 minute, contrast free MRI scan that provides three metrics on liver health namely fat, iron and fibro-inflammatory scores

SUMMARY:
The primary aim of this study is to investigate whether the baseline cT1 can predict those whose condition relapses following treatment withdrawal.

The secondary aim is to investigate correlation of cT1 with histology to explore utility as a monitoring tool.

A total of 97 patients with AIH will be recruited and divided into 2 arms. 20 of which will be treatment naive and the other 77 will have been on treatment for the past 18-24 months and will be coming in for therapy cessation review.

DETAILED DESCRIPTION:
Patients with AIH who have been undergoing immunosuppressive treatment for 18-24 months will be invited for a series of multiparametric MRI (mpMRI) scans to assess the utility of LMS for monitoring characteristics of the disease.

This will be a prospective, cross-sectional, observational study recruiting 97 participants (20 of which will be treatment naïve at recruitment) from those patients scheduled for a liver biopsy for therapy cessation review. They will be consented and invited for a LiverMultiScan.

All patients whose treatment is ended based on histology results will be followed up over the subsequent 12 months, and those that experience a biochemical relapse or 'flare-up' will be invited for a second LiverMultiScan prior to their scheduled liver biopsy.

All participants will attend their planned outpatient hepatology appointment with their doctor, who will document the intended treatment plan for each participant in line with their usual care pathway. Their MRI scan will then be scheduled for the same day as their outpatient appointment or within a 7-day window after their appointment with the consultant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing management for AIH being considered for treatment cessation
* Patients diagnosed with AIH, are treatment naïve, and will be undergoing biopsy as per clinical pathway
* Diagnostic biopsy prior to cessation of treatment (where possible)
* 18+ years of age.
* Ability to give informed consent

Exclusion Criteria:

* Any contraindication to MRI scanning
* Any clinically significant medical or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To assess the utility of cT1 to risk stratify patients with Autoimmune Hepatitis (AIH)
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
To assess the utility of cT1 to risk stratify patients with Autoimmune Hepatitis (AIH). | 36 months
  Performance of cT1, as assessed by Area Under the Receiver Operating Curve, for predicting those patients likely to relapse following treatment cessation.

SECONDARY OUTCOMES:
To assess the utility of cT1 to monitor active disease along the clinical pathway | 36 months
  Performance of cT1 to predict active disease, as defined by histology and assessed by Area Under the Receiver Operating Curve, as part of the monitoring pathway
To assess the correlation between cT1 and other clinically relevant outcomes and biomarkers such as blood biomarkers, autoimmune markers, ultrasound, histology and patient-reported outcome measures | 36 months
  Correlation between cT1 and other clinically relevant outcomes and biomarkers used in the AIH pathway (LFTs, autoimmune markers, ultrasound, histology and patient reported outcome measures)
To collect health economic information about adding LMS into standard care pathway | 36 months
  To quantify the potential reduction in patient management costs by reducing unnecessary appointments

CONTACTS AND LOCATIONS:
Locations (1):
- Touchstone Medical Imaging, Fort Worth, Texas, United States